CLINICAL TRIAL: NCT05022316
Title: COHERE - COntextualized Care in cHcs' Electronic Health REcords
Acronym: COHERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: OCHIN, Inc. (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01MD014886 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
Keywords: Social Determinants of Health; Decision Support Systems, Clinical; Electronic Health Records; Community Health Centers; Health Status Disparities
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A randomized quasi-experimental design will be used to assess the impact of the newly developed CDS tools designed to support social-risk informed care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Control clinics will not receive an intervention.
- Intervention Arm (Experimental): Intervention clinics will have the CDS tools turned on in their EHR.
  Interventions: Other: CDS Tool Access

INTERVENTIONS:
Other: CDS Tool Access — Clinics receiving the intervention will have access to EHR-based CDS tools designed to support social risk-informed care. Prior to tool activation in participating community health centers (CHCs), clinic staff members will be oriented to the CDS tools by an EHR trainer (either on-site or remotely).
  Arms: Intervention Arm

SUMMARY:
This study was designed to develop and test clinical decision support (CDS) tools that present clinical care team members with a given patient's social risk information and recommend care plan adaptations based on those risks. This study will test the hypothesis that providing care team members with CDS about patients' known social risks will result in improved outcomes. This study's primary outcomes are hypertension and diabetes control, but the results will have implications for a wide range of morbidities.

DETAILED DESCRIPTION:
The investigators will use a randomized quasi-experimental design to assess impact of the CDS tools designed to support social risk-informed care. After conducting a 12-month pilot study with 3 CHCs to test and further refine the CDS tools, 6 CHCs will be recruited to participate in the main trial. All OCHIN clinics with >200 SDH screenings (excluding the pilot clinics) will be identified and randomized to a potential intervention group or a control group. Clinics from the potential intervention group will be recruited in a random order until 6 agree to participate. This recruitment method ensures randomization between intervention and control clinics, without recruiting CHCs to a study in which they might not receive an intervention. Intervention sites will be trained in how to use the tools shortly before the tools are activated and will be followed for 12 months to assess tool adoption and impact on the CQMs of interest. Use of the CDS tools will occur as part of the regular care patients receive and will not require special clinic visits. Patients will interact with providers as they normally would, augmented by the intervention when clinicians choose to utilize the CDS tools. For all study clinics, quantitative data will be collected (via EHR data extraction) on social risk data collection and action by care team members. Limited clinical data will be collected on patients who are seen at a study CHC during the study period. Qualitative data will also be collected which includes semi-structured interviews with clinic staff from all study CHCs enrolled in the main trial.

NOTE: Individual patients will not be assigned to an intervention. Instead, randomization and intervention will occur at the clinic level. While CHCs will be recruited that have previously screened patients for social risks, it is unlikely that these CHCs will have screened all patients in their clinics. Thus, the CDS tools will not apply to all patients in participating clinics, and it cannot be guaranteed that individual patients will receive an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinic has conducted >200 social risk screenings in the last 12 months at the time of randomization.
* Clinic provides primary care
* Joined OCHIN by 07/01/2021

Exclusion Criteria:

* Clinic participated in pilot
* Clinic is a school-based health center
* Clinic provides care to prison population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
hypertension control | 12 months
  binary outcome of patient having a blood pressure of <140/90 at the time of the clinic visit (0=no, 1=yes)
diabetes control | 12 months
  binary outcome of patient with diabetes having an HbA1c of <9% at the time of the clinic visit (0=no, 1=yes)

SECONDARY OUTCOMES:
completion of social risk screening | 12 months
  binary outcome of patient whose last social risk screening is >12 months old at the time of an encounter (0=no, 1=yes)
SDH z-codes added to problem list and/or visit list | 12 months
  binary outcome of patient with a positive screening for social risks and without an associated SDH z-code having the z-code added to the problem/visit list (0=no, 1=yes)
completion of medication adherence documentation | 12 months
  binary outcome of patient with prescribed medications has up-to-date medication adherence data documented in the EHR (0=no, 1=yes)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gold, PhD, MPH, Principal Investigator — Kaiser Permanente Center for Health Research; OCHIN; Laura Gottlieb, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - OCHIN, Inc, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
All EHR data are proprietary to the OCHIN clinics and thus will not be made directly available beyond the study team.

REFERENCES:
- [Derived] Gunn R, Pisciotta M, Gold R, Bunce A, Dambrun K, Cottrell EK, Hessler D, Middendorf M, Alvarez M, Giles L, Gottlieb LM. Partner-developed electronic health record tools to facilitate social risk-informed care planning. J Am Med Inform Assoc. 2023 Apr 19;30(5):869-877. doi: 10.1093/jamia/ocad010. PMID 36779911